CLINICAL TRIAL: NCT01479400
Title: Safety Study for Infants Who Exposed to Antipsychotics as Fetus
Brief Title: Effects of Exposed to Antipsychotics Throughout Pregnancy on Infants Development: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, primary investigator, Central South University
Other Study IDs: WU30971052
Record Dates: First submitted 2011-11-16; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Schizophrenia
Keywords: antipsychotic; schizophrenia; infant development
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- infants who were exposed to antipsychotics as fetus
- infants who were not exposed to antipsychotics as fetus

SUMMARY:
The primary aim of this prospective study is to evaluate the effect of antipsychotics on infant development especially neurobehavioral development which evaluated by the Bayley-III when mothers are treated with antipsychotics throughout their pregnancy.

DETAILED DESCRIPTION:
The neurodevelopmental effect of antipsychotics on fetus has always been a major concern for women who need antipsychotic treatments and are in their reproductive years. The fear of harmful effects from antipsychotic on fetus and unplanned pregnancy commonly causes non-adherence to treatments. Even for those who are willing to maintain their antipsychotic treatments during pregnancy, the fear of potential harmful effects from antipsychotic on fetus can still exist. It is well known that non-adherence to antipsychotic treatments in patients with schizophrenia can cause most to relapse and poor treatment response. The consequences of relapse not only increase personal suffering, but also increase family and societal burden.Clearly, it is important to evaluate the safety of antipsychotics during pregnancy. However, up to now, most information about antipsychotics on reproductive safety and the effects on infant development come from case reports, case series, and retrospective studies.So the study was to investigate the developmental effects of antipsychotics on infants who were exposed to as fetus.

ELIGIBILITY:
Inclusion Criteria:

* newborns
* exposed to antipsychotic as fetus
* no exposed to antipsychotic

Exclusion Criteria:

* malformation
* liver dysfunction
* renal dysfunction
* cardiovascular diseases

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 76 infants who were exposed to antipsychotics as fetus was compared to 76 matched control infants who were not exposed to antipsychotics as fetus.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
evidence of negative effects of antipsychotic on infant mental development confirmed by Bayley Scales of Infant and Toddler Development | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute, Changsha, Hunan, China

REFERENCES:
- [Derived] Shao P, Ou J, Peng M, Zhao J, Chen J, Wu R. Effects of Clozapine and other Atypical Antipsychotics on Infants Development Who Were Exposed to as Fetus: A Post-Hoc Analysis. PLoS One. 2015 Apr 24;10(4):e0123373. doi: 10.1371/journal.pone.0123373. eCollection 2015. PMID 25909513
- [Derived] Peng M, Gao K, Ding Y, Ou J, Calabrese JR, Wu R, Zhao J. Effects of prenatal exposure to atypical antipsychotics on postnatal development and growth of infants: a case-controlled, prospective study. Psychopharmacology (Berl). 2013 Aug;228(4):577-84. doi: 10.1007/s00213-013-3060-6. Epub 2013 Apr 5. PMID 23559219